CLINICAL TRIAL: NCT02898805
Title: Effects of a New Combination of Nutraceutics (LopiGLIK®) on Cardiovascular Risk
Brief Title: Effects of LopiGLIK® on Cardiovascular Risk
Acronym: LopiWEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, PROF OF CARDIOLOGY, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AKP_3
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Risk Factors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LopiGLIK® (Experimental): first two weeks: Placebo + prescribed Diet then 16 weeks LopiGLIK® a tablet/day after a meal + Diet
  Interventions: Other: Placebo; Other: Prescribed Diet; Dietary Supplement: LopiGLIK®
- Armolipid Plus (Active Comparator): first two weeks: Placebo + prescribed Diet then 16 weeks Armolipid Plus a tablet/day after a meal + Diet
  Interventions: Other: Placebo; Other: Prescribed Diet; Dietary Supplement: Armolipid Plus

INTERVENTIONS:
Other: Placebo
Other: Prescribed Diet
Dietary Supplement: LopiGLIK®
  Arms: LopiGLIK®
Dietary Supplement: Armolipid Plus
  Arms: Armolipid Plus

SUMMARY:
The study is designed to compare the effects of two combination of nutraceuticals: Armolipid Plus® and LopiGLIK® (Akademy Pharma), a new supplement that, in addition to Berberine and Red Rice, contains Morus Alba's extract. The study will analyze the impact of 16 week treatment with one of the combinations, according to a randomized scheme, on metabolic parameters in dyslipidemic subjects that do not require or not tolerate a statin therapy. In particular, it will assess the ability of the two combinations to reduce the levels of total and LDL cholesterol, HbA1C, glicaemia and insulin and increase those of HDL cholesterol.

DETAILED DESCRIPTION:
The experimental design involves the construction of a multi-center, controlled, randomized, single-blind, versus Armolipid Plus®.

Patients with mild hypercholesterolemia, of both sexes and aged between 18 and 75 years, will be recruited, from the beginning of the study and for the next 2 weeks, from 30 Cv specialists and/or GPs (25 patients each).

The subjects will be enrolled in the 50/50% male/female ratio ± 10% comparable for age, in order to obtain a proper comparison between groups with similar demographic characteristics or not statistically different.

The subjects, selected on the basis of inclusion and exclusion criteria, will be divided into two groups, subjected to centralized randomization at the "Diagnosis and Treatment of hypertension Center" to receive one of two different treatments, a tablet/day of the new nutraceutical LopiGLIK® (Akademy Pharma) containing Morus Alba, immediately after a meal, vs. a tablet/day of Armolipid Plus, always immediately after the meal. During the first two weeks both groups will follow the prescribed diet and assume the placebo. At the end, blood tests (traditional metabolic parameters, blood glucose, HbA1C, fasting insulin, transaminase levels, CPK) and the endothelial function will be assesed. During the next 16 weeks a group will assume LopiGLIK® (Akademy Pharma) containing Morus Alba, the other will assume Armolipid Plus and everyone will continue to follow the prescribed diet. At the end of this period blood tests will be repeated. Tablets of Armolipid Plus, LopiGLIK® and placebo will be provided by Akademy Pharma free of charge

ELIGIBILITY:
Inclusion Criteria:

* Total Cholesterol<300 mg/dL
* Total Cholesterol>200 mg/dL
* Cardiovascular Risk<20%

Exclusion Criteria:

* Pregnancy
* Documented intolerance to one or more 'components LOPIGLIK / Armolipid PLUS
* Previous cardiovascular events
* Familiar severe dyslipidemia
* Familiar high cardiovascular risk Hepatic or muscular disorders Subjects receiving lipid-lowering drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Reduction of LDL-Cholesterol levels | 16 weeks

SECONDARY OUTCOMES:
Increasing of HDL-Cholesterol levels | 16 weeks
Reduction of HbA1c levels | 16 weeks
Reduction of fastin insuline levels | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, Professor, Principal Investigator — FEDERICO II UNIVERSITY - NAPLES
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data available to principal investigator

REFERENCES:
- [Result] Trimarco V, Izzo R, Stabile E, Rozza F, Santoro M, Manzi MV, Serino F, Schiattarella GG, Esposito G, Trimarco B. Effects of a new combination of nutraceuticals with Morus alba on lipid profile, insulin sensitivity and endotelial function in dyslipidemic subjects. A cross-over, randomized, double-blind trial. High Blood Press Cardiovasc Prev. 2015 Jun;22(2):149-54. doi: 10.1007/s40292-015-0087-2. Epub 2015 Apr 14. PMID 25870124
- [Result] Carrizzo A, Ambrosio M, Damato A, Madonna M, Storto M, Capocci L, Campiglia P, Sommella E, Trimarco V, Rozza F, Izzo R, Puca AA, Vecchione C. Morus alba extract modulates blood pressure homeostasis through eNOS signaling. Mol Nutr Food Res. 2016 Oct;60(10):2304-2311. doi: 10.1002/mnfr.201600233. Epub 2016 Jun 27. PMID 27234065
- [Derived] Manfrin A, Trimarco V, Manzi MV, Rozza F, Izzo R. A single blind, multicenter, randomized controlled trial to evaluate the effectiveness and cost of a novel nutraceutical (LopiGLIK(R)) lowering cardiovascular disease risk. Clinicoecon Outcomes Res. 2018 Oct 8;10:601-609. doi: 10.2147/CEOR.S172838. eCollection 2018. PMID 30349338